CLINICAL TRIAL: NCT00324272
Title: Can Fibrin Sealant be Used to Reduce Post-operative Drainage Following Lymph Node Dissection: a Prospective Randomised Double Blind Trial.
Brief Title: Post-Operative Drainage Following Lymph Node Dissection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Mr. H. Giele, Consultant Plastic & Reconstructive Surgeon, Oxford Radcliffe Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C02.240
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2006-05

CONDITIONS: Malignant Melanoma; Carcinoma, Squamous Cell
Keywords: Groin dissection; Axilla (or axillary) dissection; Lymph node dissection; Lymphadenectomy; Seroma; Wound drainage; Fibrin sealant; Malignant melanoma; Squamous cell carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Squamous Cell; Seroma | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Groin dissection: sealant used. (Experimental)
  Interventions: Drug: Fibrin Sealant (Tisseel) used in the Experimental Arm.
- Groin dissection: no sealant used. (Active Comparator)
  Interventions: Drug: Fibrin Sealant (Tisseel) used in the Experimental Arm.
- Axillary dissection: sealant used. (Experimental)
  Interventions: Drug: Fibrin Sealant (Tisseel) used in the Experimental Arm.
- Axillary dissection: no sealant used. (Active Comparator)
  Interventions: Drug: Fibrin Sealant (Tisseel) used in the Experimental Arm.

INTERVENTIONS:
Drug: Fibrin Sealant (Tisseel) used in the Experimental Arm. — For patients in the Experimental (Treatment) Arm, 4 ml of Tisseel fibrin sealant were instilled into the wound using the Duploject™ spray delivery system prior to wound closure. Tisseel™ fibrin sealant was provided by Baxter Healthcare Ltd., Newbury, Berkshire, UK.
  For patients in the Active Comparator (Control) Arm, no fibrin sealant was used during wound closure (with the surgical procedure being identical in all other respects).

SUMMARY:
The purpose of this study is to determine whether the use of fibrin sealant reduces post-operative drainage following groin and axillary lymph node dissection.

DETAILED DESCRIPTION:
Background: Fibrin sealant has been used for many years in clinical practice and has a wide range of applications including the control of lymphatic leaks and haemostasis. The physiological mechanism of action of fibrin was first described by Morawitz in 1905; fibrin sealant was first marketed in 1983.

Lymph node dissection is undertaken for the control of malignant disease - frequently malignant melanoma or squamous cell carcinoma. Following groin or axillary dissection, excessive post operative drainage may necessitate the presence of wound drains for 10 days or more. This may prolong hospital stay in some patients, and may be associated with an increased complication rate (such as wound infection).

Hypothesis: the use of fibrin sealant prior to wound closure following either groin or axillary dissection may reduce post-operative wound drainage.

Comparison: patients who require an elective groin or axillary dissection who either undergo standard wound closure or those who have fibrin sealant instilled into the surgical wound prior to wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Requiring groin or axillary lymph node dissection for malignant disease.

Exclusion Criteria:

* Patients under age 18 years.
* Patients unable to speak English.
* Patients with learning difficulties.
* Patients with mental illness.
* Prisoners.
* Other vulnerable groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-01; Primary Completion 2006-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henk P. Giele, MBBS FRACS, Principal Investigator — UK: National Health Service

REFERENCES:
- [Background] Oliver DW, Hamilton SA, Figle AA, Wood SH, Lamberty BG. A prospective, randomized, double-blind trial of the use of fibrin sealant for face lifts. Plast Reconstr Surg. 2001 Dec;108(7):2101-5, discussion 2106-7. doi: 10.1097/00006534-200112000-00044. PMID 11743409
- [Background] Moore MM, Nguyen DH, Spotnitz WD. Fibrin sealant reduces serous drainage and allows for earlier drain removal after axillary dissection: a randomized prospective trial. Am Surg. 1997 Jan;63(1):97-102. PMID 8985079
- [Background] Berger A, Tempfer C, Hartmann B, Kornprat P, Rossmann A, Neuwirth G, Tulusan A, Kubista E. Sealing of postoperative axillary leakage after axillary lymphadenectomy using a fibrin glue coated collagen patch: a prospective randomised study. Breast Cancer Res Treat. 2001 May;67(1):9-14. doi: 10.1023/a:1010671209279. PMID 11518470
- [Background] Giovannacci L, Renggli JC, Eugster T, Stierli P, Hess P, Gurke L. Reduction of groin lymphatic complications by application of fibrin glue: preliminary results of a randomized study. Ann Vasc Surg. 2001 Mar;15(2):182-5. doi: 10.1007/s100160010049. Epub 2001 Mar 1. PMID 11265082
- [Background] Jain PK, Sowdi R, Anderson AD, MacFie J. Randomized clinical trial investigating the use of drains and fibrin sealant following surgery for breast cancer. Br J Surg. 2004 Jan;91(1):54-60. doi: 10.1002/bjs.4435. PMID 14716794
- [Result] Swan MC, Oliver DW, Cassell OC, Coleman DJ, Williams N, Morritt DG, Giele HP. Randomized controlled trial of fibrin sealant to reduce postoperative drainage following elective lymph node dissection. Br J Surg. 2011 Jul;98(7):918-24. doi: 10.1002/bjs.7462. Epub 2011 Apr 1. PMID 21456091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred between 1.1.2003 and 31.12.2006. A total of 74 patients were recruited. All patients were followed up until 1.6.2010.
Pre-assignment Details: All 74 patients who were enrolled in the trial were followed up until 1.6.10 (unless they died prior to this date).
Groups:
- Groin Dissection: Sealant Used.: All infrainguinal nodes, including Cloquet's node, were removed in all groin dissection cases. Routine peri-operative antibiotic prophylaxis was used. Diathermy and ligating clips were used as required and the wound bed irrigated with sterile water prior to closure. Closed suction drains were inserted and secured with drain sutures. 4 ml of Tisseel fibrin sealant (containing 1000 IU of human thrombin as the 'fast-set' preparation) were instilled into the wound using the Duploject™ spray delivery system. Firm pressure was applied to the wound for three minutes whilst the sealant set in order to obliterate the dead space, following which the skin was closed in two layers using absorbable sutures and the drains were vacuumed. A dry dressing was applied.
- Groin Dissection: no Sealant Used.: All infrainguinal nodes, including Cloquet's node, were removed in groin dissection cases. Routine peri-operative antibiotic prophylaxis was used. Diathermy and ligating clips were used as required and the wound bed irrigated with sterile water prior to closure. Closed suction drains were inserted and secured with drain sutures. No Tisseel fibrin sealant was instilled into the wound. The skin was closed in two layers using absorbable sutures and the drains were vacuumed. A dry dressing was applied.
- Axillary Dissection: Sealant Used.: A level I to III nodal clearance was performed in axillary dissection cases. Routine peri-operative antibiotic prophylaxis was used. Diathermy and ligating clips were used as required and the wound bed irrigated with sterile water prior to closure. Closed suction drains were inserted and secured with drain sutures. 4 ml of Tisseel fibrin sealant (containing 1000 IU of human thrombin as the 'fast-set' preparation) were instilled into the wound using the Duploject™ spray delivery system. Firm pressure was applied to the wound for three minutes whilst the sealant set in order to obliterate the dead space, following which the skin was closed in two layers using absorbable sutures and the drains were vacuumed. A dry dressing was applied.
- Axillary Dissection: no Sealant Used.: A level I to III nodal clearance was performed in axillary dissection cases. Routine peri-operative antibiotic prophylaxis was used. Diathermy and ligating clips were used as required and the wound bed irrigated with sterile water prior to closure. Closed suction drains were inserted and secured with drain sutures. No Tisseel fibrin sealant was instilled into the wound. The skin was closed in two layers using absorbable sutures and the drains were vacuumed. A dry dressing was applied.
Period: Overall Study
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Started | 18 | 20 | 18 | 18
Completed | 18 | 20 | 18 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used. | Total
Number analyzed (Participants) | 18 | 20 | 18 | 18 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 10 | 16 | 51
  >=65 years | 6 | 7 | 8 | 2 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (17.9) | 58.2 (18.1) | 64.7 (18.4) | 57.3 (14.2) | 58.1 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 7 | 6 | 35
  Male | 9 | 7 | 11 | 12 | 39
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18 | 20 | 18 | 18 | 74

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Wound Drainage.
Description: The postoperative wound drainage volume was measured from the day of surgery until the the date of removal of the last wound drain.
Time Frame: From date of surgery to date of wound drain removal (typically a period of approximately one week).
Measure: Median (95% Confidence Interval); unit: ml
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 18 | 20 | 18 | 18
ml | 892.5 [265 to 2895] | 762.5 [25 to 3255] | 565 [30 to 1835] | 590 [230 to 9605]
Statistical Analysis 1: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.704, t-test, 2 sided
Statistical Analysis 2: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.217, t-test, 2 sided

2. Secondary Outcome: Length of Hospital Inpatient Stay.
Description: The length of hospital stay was calculated from the day of surgery to the day that the patient was discharged from hospital.
Time Frame: From date of surgery until date of discharge from hospital.
Population: As the length of hospital stay was affected by numerous factors other than those related to the surgery itself (e.g. the patient's social circumstances), the results for this secondary outcome measure have not been presented.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Length of Time Drains Remain in Situ.
Description: The duration of postoperative wound drainage was measured from the day of surgery until the the date of removal of the last wound drain.
Time Frame: From date of surgery until date of wound drain removal.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 18 | 20 | 18 | 18
Days | 7 [5 to 15] | 7.5 [2 to 37] | 7.5 [1 to 15] | 9 [3 to 26]
Statistical Analysis 1: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.988, t-test, 2 sided
Statistical Analysis 2: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.426, t-test, 2 sided

4. Secondary Outcome: Number of Patients With Post-operative Complications (Excluding Lymphoedema).
Description: Complications were classified as being either 'Minor' (i.e. (managed without operation, prolonged hospital stay or readmission) or 'Major' (i.e. requiring surgical intervention or readmission to hospital). The number of patients with each 'Minor' and 'Major' complication were recorded.
Time Frame: Until wound healing complete.
Measure: Number; unit: Participants
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 18 | 20 | 18 | 18
Participants | 12 | 16 | 13 | 12
Statistical Analysis 1: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.351, Fisher Exact
Statistical Analysis 2: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.480, Fisher Exact

5. Secondary Outcome: Post Operative Pain Score Measured on 1st Post-operative Day.
Description: Pain score was recorded at 24 hours following the completion of surgery using a Visual Analogue Score (using a scale of 1 [no pain] to 10 [very severe pain]) which the patient was asked to record.
Time Frame: During the immediate post-operative period.
Measure: Median (Inter-Quartile Range); unit: Units on a scale.
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 18 | 20 | 18 | 18
Units on a scale. | 1 [1 to 1.25] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 2]
Statistical Analysis 1: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Test type: Superiority or Other; p = 0.400, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Disease Recurrence.
Description: This was measured as either: 1. the number of participants with local recurrence; 2. the number of participants with in transit or regional recurrence; or 3. the number of participants with distant metastasis (but alive on 1st June 2010).
Time Frame: From date of surgery until end of study follow-up period (1st June 2010)
Measure: Number; unit: Participants.
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 18 | 20 | 18 | 18
Participants. | 11 | 6 | 5 | 8
Statistical Analysis 1: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Local recurrence in the groin cohort; Test type: Superiority or Other; p = 1.00, Fisher Exact
Statistical Analysis 2: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; In transit or regional recurrence in the groin cohort; Test type: Superiority or Other; p = 0.301, Fisher Exact
Statistical Analysis 3: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Distant metastasis in the groin cohort (with the patient being alive at the end of the study follow-up period on 1.6.10); Test type: Superiority or Other; p = 0.474, Fisher Exact
Statistical Analysis 4: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Local recurrence in the groin cohort; Test type: Superiority or Other; p = 0.606, Fisher Exact
Statistical Analysis 5: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; In transit or regional recurrence in the axillary cohort; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 6: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Distant metastasis in the axillary cohort (with the patient being alive at the end of the study follow-up period on 1.6.10); Test type: Superiority or Other; p = 0.486, Fisher Exact

7. Secondary Outcome: Death.
Description: Death was recorded as the number of participants who had died by the end of the study follow-up period (1st June 2010). Deaths were recorded as either being related to the primary disease (i.e. due to distant metastasis) or death due to another (unrelated) cause (e.g. myocardial infarction or cerebrovascular accident).
Time Frame: From day of surgery until end of study follow-up period (1st June 2010)
Measure: Number; unit: Participants.
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Number analyzed (Participants) | 18 | 20 | 18 | 18
Participants. | 10 | 12 | 9 | 9
Statistical Analysis 1: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Death from metastatic disease in the groin cohort; Test type: Superiority or Other; p = 0.963, Regression, Cox; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.40 to 2.58]
Statistical Analysis 2: Comparison: Groin Dissection: Sealant Used. vs Groin Dissection: no Sealant Used; Death from an unrelated cause in the groin cohort; Test type: Superiority or Other; p = 0.338, Regression, Cox; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.03 to 3.20]
Statistical Analysis 3: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Death from metastatic disease in the axillary cohort; Test type: Superiority or Other; p = 0.880, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.35 to 2.47]
Statistical Analysis 4: Comparison: Axillary Dissection: Sealant Used. vs Axillary Dissection: no Sealant Used; Death from an unrelated cause in the axillary cohort; Test type: Superiority or Other; p = 0.923, Regression, Cox; Hazard Ratio (HR) = 0.923, 95% CI 2-sided [0.05 to 13.95]

ADVERSE EVENTS:
Time Frame: From date of surgery (i.e. date of randomization) until the date of the adverse event (e.g. death, seroma formation) or the end of study follow-up period (1st June 2010) whichever is the sooner.
Arm/Group | Groin Dissection: Sealant Used. | Groin Dissection: no Sealant Used. | Axillary Dissection: Sealant Used. | Axillary Dissection: no Sealant Used.
Serious Adverse Events (participants affected / at risk) | 10/18 | 12/20 | 9/18 | 9/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Groin Dissection: Sealant Used. (N=18) | Groin Dissection: no Sealant Used. (N=20) | Axillary Dissection: Sealant Used. (N=18) | Axillary Dissection: no Sealant Used. (N=18)
Death (General disorders) | 10 (10) | 12 (12) | 9 (9) | 9 (9)
Wound Seroma (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 5 (5) | 5 (5) — Non-infected post-operative seroma requiring outpatient aspiration. In this category the seroma is neither infected nor does it require inpatient treatment (e.g. surgical drainage).
Wound cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Wound necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Infected seroma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) — Infected post-operative seroma requiring admission for intravenous antibiotics but not requiring surgical drainage.
Surgical seroma (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6) | 3 (3) | 0 (0) — Infected post-operative seroma requiring admission to hospital for incision & drainage procedure.
Haematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Post-operative haematoma requiring surgical drainage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes